CLINICAL TRIAL: NCT03929653
Title: Prospective and Retrospective Register Study of Personalized Therapy of Molecular Tumor Board Participation With The Guidance of Next Generation Sequencing
Brief Title: Personalized Therapy of Molecular Tumor Board Participation With the Guidance of Next Generation Sequencing
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MTB-PT
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Solid Tumor, Adult
Keywords: Next Generation Sequencing; Personalized Therapy; Molecular Tumor Board
MeSH Terms: interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Refractory Solid Tumors: Patients with advanced refractory solid tumors receive personalized therapy with the guidance of Molecular Tumor Board after the NGS(next generation sequencing).
  Interventions: Other: Personalized therapy model with Molecular Tumor Board and Next Generation Sequencing

INTERVENTIONS:
Other: Personalized therapy model with Molecular Tumor Board and Next Generation Sequencing — This study is to observe this therapy model outcomes

SUMMARY:
This study seeks to evaluate the clinical value of the personalized therapy model with the guidance of Molecular Tumor Board (MTB) after Next Generation Sequencing(NGS), and to track patient outcomes.

DETAILED DESCRIPTION:
This is a study from the real world. Advanced refractory solid tumors patients with no standard treatment options have a very poor prognosis. In recent years, the application of s Next Generation Sequencing (NGS) has rapidly expanded the breadth and depth of understanding of the molecular mechanism of tumors, laying a foundation for the development of precision medicine for tumors. Researchers can build a molecular phenotype of advanced refractory solid tumors by NGS. Some retrospective study shows that Molecular Tumor Board (MTB) therapy model brings therapeutic hope. So, investigators hope that this therapy model combined with NGS may provide treatment recommendations for advanced refractory solid tumors patients. Those recommendations may include some off-label targeted therapies. This study seeks to evaluate the clinical value of the personalized therapy model with the guidance of MTB after NGS, and to track patient outcomes, including ORR (Objective Response Rate), PFS (Progression Free Survival), OS (Overall Survival) and ADR (Adverse Drug Reaction).

ELIGIBILITY:
Inclusion Criteria:

1. Is equal to or greater than 18 years of age.
2. Histologic or cytologic confirmation of advanced refractory solid tumors with no standard treatment options, including some patients with advanced disease in reduced general condition (Eastern Cooperative Oncology Group (ECOG) 3 and 4).
3. Patients with measurable or evaluable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
4. Patients must be able to provide blood samples or tissue samples for NGS (Next Generation Sequencing) testing. The amount of blood and tissue samples should be able to meet the requirements of DNA extraction and quality control.
5. Adequate baseline organ system function.
6. Patients could receive treatment program from MTB (Molecular Tumor Board).
7. Ability to understand and the willingness to provide a written informed consent document.

Exclusion Criteria:

1.According to the investigator' judgment, there are serious, uncontrollable risks to patients' safety, or associated diseases (such as severe diabetes, thyroid disease, infection, spinal cord compression, superior vena cava syndrome, neurological or psychiatric disorders and so on) that affect the patients completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The objective is to describe in a real-world advanced refractory solid tumors population. First of all, this study will be carried out as a retrospective, observational review of patients who clinically diagnosed as advanced refractory solid tumors received personalized therapy with the guidance of MTB (molecular tumor board) after the NGS (next generation sequencing). Then, the investigators prospective observation personalized therapy plan which the MTB recommends for patients who clinically diagnosed as advanced refractory solid tumors according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective Response Rate) | Up to three months
  ORR is the percentage of participants with best overall response of complete response (CR), partial response (PR). Response categories: CR, PR, SD (stable disease), PD (progressive disease) Criteria on which physicians determined therapy response also will be captured by using Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 to evaluate.

SECONDARY OUTCOMES:
PFS (Progression Free Survival), calculated from various time points | Up to two years
  Progression-free survival (PFS) is defined as progression free survival of all the evaluable participants who receive targeted drug therapy. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1).
OS (Overall Survival), calculated from various time points | Duration of time from the start of treatment to date of death, assessed up to 2 years
  OS is defined as time from initiation to death of any cause.
ADR (Adverse Drug Reaction) | 30 days after last dose.
  Adverse events determined according to CTCAE (version 4.03).

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Principal Investigator — Tianjin Medical Unversity Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided